CLINICAL TRIAL: NCT06373718
Title: A Novel Use of a Sleep Intervention to Target the Emotion Regulation Brain Network to Treat Depression and Anxiety (R33 Phase)
Brief Title: Sleep Mechanisms Of Regulating Emotions
Acronym: SleepMORE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Andrea Goldstein-Piekarski, Assistant Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-74553; R33MH120245 (NIH)
Record Dates: First submitted 2024-04-15; First posted 2024-04-18 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Insomnia; Depression
Keywords: Insomnia; Depression; Anxiety; CBT-I; Cognitive Behavioral Therapy for Insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Depression; Anxiety Disorders | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be randomized into either the Immediate Treatment group, or the Enhanced Sleep Hygiene group. Both study groups will receive CBT-I.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Treatment (Experimental): Participants randomized to the Immediate Treatment group will receive CBT-I treatment immediately after randomization.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia
- Enhanced Sleep Hygiene (Other): Participants randomized to the Enhanced Sleep Hygiene (ESH) group will be offered the same CBT-I described above approximately 7 months after being randomized. We will also provide a list of referrals for treatment upon completion of their end of treatment visit (approx. week 11) should they choose to seek treatment sooner. In the interim, they will be provided with two sessions of sleep hygiene / sleep education and four additional meetings including monitoring of sleep and mood symptoms.
  Interventions: Behavioral: Cognitive Behavioral Therapy for Insomnia

INTERVENTIONS:
Behavioral: Cognitive Behavioral Therapy for Insomnia — CBT-I improves sleep through a combination of behavioral interventions (stimulus control (SC), sleep restriction (SR)), cognitive therapy (CT) as well as additional components such as mindfulness training and sleep hygiene education. SC is an intervention that re-establishes the connection between the bed/bedroom with sleep to help develop a more consistent sleep/wake pattern. SR leads to higher quality sleep by reducing excessive time spent in bed to the actual amount of sleep, thereby creating mild sleep deprivation and increasing the homeostatic sleep drive. Like CT for other disorders, CT for insomnia targets maladaptive thoughts and cognitions that may interfere with sleep.
  Other Names: CBT-I

SUMMARY:
This project is the second phase of a two-phased project investigating the impact of a proven sleep intervention, Cognitive Behavioral Therapy for Insomnia (CBT-I) on engagement of the emotion regulation brain network as a putative mechanistic target.

DETAILED DESCRIPTION:
Several lines of evidence suggest that insomnia contributes to emotionally distressing depressive mood symptoms through disruption of brain networks that regulate emotional functions. Of particular concern, insomnia is associated with an increased risk for suicide, even when accounting for the presence of other depressive symptoms. However, it is not yet know to what degree that the emotion regulation brain network is modified by the restoration of sleep, or whether the degree to which a sleep intervention engages these neural targets mediates reductions in depressive symptoms and suicidality.

This project is the second phase of a two-phased project investigating the impact of a proven sleep intervention, Cognitive Behavioral Therapy for Insomnia (CBT-I) on engagement of the emotion regulation brain network as a putative mechanistic target.

This project aims to extend the initial findings from the first phase (IRB-56961) to (1) confirm target engagement, defined as the treatment effect on increasing mPFC-amygdala connectivity, and/or decreasing amygdala reactivity during emotion reactivity and regulation paradigms, by testing the hypothesis that compared with a control condition, CBT-I participants will show significant change in the emotion regulation network targets that met the Go Criteria of the first phase in the direction of normalization, at the end of treatment, (2) examine the relationships of target engagement to treatment outcomes by study group, and (3) test whether emotion regulation network measures at baseline predict depressive symptom and suicidality reduction.

Participants will be 150 adults experiencing at least moderate sleep disturbances and who also have elevated anxious and/or depressive symptoms. Eligible participants will be randomized into either the Immediate Treatment group, which will receive six sessions of CBT-I over the eight weeks of treatment phase immediately after randomization, or the Enhanced Sleep Hygiene group, which will be provided with two sessions of sleep hygiene / sleep education and four additional meetings including monitoring of sleep and mood symptoms and will be offered the same CBT-I as the Immediate Treatment group upon completion of the 6-month follow-up session, approximately 7 months after randomization. Emotion distress and sleep disruption will be assessed prior to, and weekly during the eight weeks of treatment phase. CBT-I improves sleep patterns through a combination of sleep restriction, stimulus control, mindfulness training, cognitive therapy targeting dysfunctional beliefs about sleep, and sleep hygiene education. Using fMRI scanning, emotion regulation network neural targets will be assayed prior to and following completion of CBT-I treatment.

ELIGIBILITY:
Inclusion Criteria:

* Males and females of any racial or ethnic group, aged 25-60
* Subjective complaint of insomnia associated with daytime impairment or distress (ISI ≥ 10)
* Insomnia complaint ≥ 3 months in duration
* Subjective complaint of depressive symptoms as defined by scores of ≥ 14 on the BDI
* Fluent and literate in English
* Written, informed consent
* Reside within 60 miles of Stanford University

Exclusion Criteria:

* Presence of other sleep or circadian rhythm disorders that significantly contribute to their sleep disturbance. The presence of these disorders will be assessed by the DUKE structured interview for sleep disorders
* Use of psychotropic medications that would significantly impact sleep, alertness, or mood and unwilling or unable to discontinue medication specifically prescribed for sleep disturbance > two weeks (anti-depressants) or >1 week (sleep medications) prior to baseline data collection
* Excessive alcohol consumption (>14 drinks per week or > 4 drinks per occasion)
* Presence of suicidal ideations representing imminent risk as determined by the empirically-supported, standardized suicide risk assessment
* General medical condition, disease or neurological disorder that interferes with the assessments
* Substance abuse or dependence
* History of significant head trauma followed by persistent neurological deficits or known structural brain abnormalities OR traumatic brain injury in the past two months
* Severe impediment to vision, hearing and/or hand movement, likely to interfere with the ability to complete the assessments, or are unable and/or unlikely to follow the study protocols
* Pregnant or breast feeding
* Current or lifetime history of bipolar disorder or psychosis
* Current or expected cognitive behavior therapy or other evidence-based psychotherapies for another condition
* Received cognitive behavioral therapy for insomnia within the past year
* Acute or unstable chronic illness: including but not limited to: uncontrolled thyroid disease, kidney, prostate or bladder conditions causing excessively frequent urination (> 3 times per night); medically unstable congestive heart failure, angina, other severe cardiac illness as defined by treatment regimen changes in the prior 3 months; stroke with serious sequelae; cancer if < 1 year since end of treatment; asthma, emphysema, or other severe respiratory diseases uncontrolled with medications; and neurological disorders such as Alzheimer's disease, Parkinson's disease and unstable epilepsy as defined by treatment regimen changes in the prior 3 months; unstable adult onset diabetes as defined by treatment regimen changes in the prior 3 months
* Current exposure to trauma, or exposure to trauma within the past 3 months
* Working a rotating shift that overlaps with 2400h
* Individuals who were high risk for sleep apnea on the Berlin Questionnaire and are not CPAP adherent or have untreated OSA of moderate severity or worse (AHI ≥ 15)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Change in Emotion Regulation Network brain activation as assessed by functional magnetic resonance imaging | Assessed at baseline (week 1) and end of treatment (week 13)
  During functional magnetic resonance imaging the Emotion Regulation Network will be engaged by emotional tasks, and circuit activation will be quantified by blood flow in regions of interest.
Change in Emotion Regulation Network brain connectivity as assessed by functional magnetic resonance imaging | Assessed at baseline (week 1) and end of treatment (week 13)
  During functional magnetic resonance imaging the Emotion Regulation Network will be engaged by emotional tasks, and circuit connectivity will be quantified by the correlation of the blood flow between regions of interest.
Change in Beck Depression Inventory | Assessed at baseline (week 1), throughout treatment phase (weeks 3-11), end of treatment (week 13), and 6-month follow-up (week 39)
  This measure is of the Beck Depression Inventory-II total score after excluding one sleep item. The average item score for the remaining 20 items will be multiplied by 21 (the original number of items), to create a modified depression scale that maintains the original range (ranges: 0-13 minimal, 14-19 mild, 20-28 moderate, and 29-63 severe).
  The BDI-II is a 21-item self-report scale with high validity and reliability that assesses the severity of depression symptoms. The depression items consist of: sadness, pessimism, past failure, loss of pleasure, guilty feelings, punishment feelings, self-dislike, self-criticalness, suicidal thoughts or wishes, crying, agitation, loss of interest, indecisiveness, worthlessness, loss of energy, irritability, changes in appetite, concentration difficulty, tiredness or fatigue, and loss of interest in sex. Items are scored from 0 to 3, and higher scores indicate greater levels of severity.
Change in PSG Sleep Efficiency | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Sleep efficiency (SE) is the percentage of total time in bed actually spent sleeping. Based on the overnight PSG sleep recording, SE will be calculated as the total time (minutes) spent asleep (sum of Stages N1, N2, N3, and REM) divided by the total time (minutes) in bed, and multiplied by 100.
Change in Insomnia Severity Index (ISI) Scale Score | Assessed at baseline (week 1), throughout treatment phase (weeks 3-11), end of treatment (week 13), and 6-month follow-up (week 39)
  Subjective ratings of sleep disturbance and insomnia severity will be assessed with the Insomnia Severity Index. The Insomnia Severity Index (ISI) is a 7-item self-report measure of insomnia type, severity, and impact on functioning. The items consist of severity of sleep onset, sleep maintenance, early morning awakenings, sleep dissatisfaction, interference with daytime functioning, noticeability of sleep problems by others, and distress caused by sleep difficulties. Items are scored from 0 to 4 (0 = no problem, 4 = very severe problem). Score ranges of insomnia are: 0-7 absent, 8-14 sub-threshold, 15-21 moderate, and 22-28 severe. The ISI has good validity and reliability.

SECONDARY OUTCOMES:
Change in Columbia Suicide Severity Rating Scale | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  The Columbia Suicide Severity Rating Scale is a 12-item checklist that was designed to quantify the severity of suicidal ideation and behavior. It is composed of two parts. The first six questions ask about suicidal ideation and behavior in the past month while the last six questions ask about suicidal ideation and behavior since the last visit. The CSSRS has been proven to be reliable and valid. It has also been shown to have high sensitivity and specificity to the different suicidal behavior classifications.
Change in Actigraph Sleep Onset Latency (SOL) as a Measure of Sleep Continuity | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Sleep Onset Latency (SOL) is the time (minutes) from "lights out" to actually falling asleep (sleep onset).
Change in Actigraph Number of Arousals as a Measure of Sleep Continuity | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Number of Arousals is determined by number of times of awakening as seen on the actigraph data.
Change in Actigraph Wake After Sleep Onset (WASO) as a Measure of Sleep Continuity | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Wake After Sleep Onset (WASO) are periods of wakefulness occurring after sleep onset, before final awakening (sleep offset).
Change in Actigraph Total Sleep Time (TST) as a Measure of Sleep Continuity | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Total Sleep Time (TST) is the total time spent asleep, from the start of sleep onset to sleep offset subtracting any periods of wakefulness.
Change in Actigraph Sleep Efficiency (SE) as a Measure of Sleep Continuity | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Sleep Efficiency (SE) is calculated as TST divided by total time spent in bed, multiplied by 100.
Change in PSG Sleep Onset Latency (SOL) as a Measure of Sleep Architecture | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Sleep Onset Latency (SOL) is the time (minutes) from "lights out" or start of total recording time, to actually falling asleep as indicated by EEG changes.
Change in PSG Number of Arousals as a Measure of Sleep Architecture | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Number of Arousals is determined by number of times of awakening by EEG changes.
Change in PSG Wake After Sleep Onset (WASO) as a Measure of Sleep Architecture | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Wake After Sleep Onset (WASO) are periods of wakefulness occurring after sleep onset, before final awakening (sleep offset) measured by EEG changes.
Change in PSG Total Sleep Time (TST) as a Measure of Sleep Architecture | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Total Sleep Time (TST) is the total time (minutes) spent asleep, from the start of sleep onset to sleep offset, subtracting any periods of wakefulness. TST includes stages N1, N2, N3, and REM sleep.
Change in PSG Sleep Efficiency (SE) as a Measure of Sleep Architecture | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Sleep Efficiency (SE) is calculated as TST divided by total time spent in bed, multiplied by 100.
  Duration of non-rapid eye movement (NREM) sleep includes stages N1, N2, and N3, and is measured in minutes. The duration of sleep outside of those stages that is associated with specific EEG stages is REM sleep.
Change in Sleep Physiology measured by PSG | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  Topographical EEG power spectral density analysis associated with sleep stages will be calculated in the Delta (0.5-Hz), Theta (4-7Hz), Alpha (7-11Hz), Sigma (12-15Hz), Beta-1 (15-20Hz), Beta-2 (20-35Hz) and Gamma (35-45Hz) bands, according to published methods.
Change in 36-Item Short Form Survey (SF-36) Score | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  The SF-36 measures health-related quality of life based on eight domains: limitations in physical activities because of health problems, limitations in social activities because of physical or emotional problems, limitations in usual role activities because of physical health problems, bodily pain, general mental health (psychological distress and well-being), limitations in usual role activities because of emotional problems, vitality (energy and fatigue), and general health perceptions. Items are recoded then averaged together to create each scale. Items that are left blank (missing data) are not taken into account when calculating the scale scores. Hence, scale scores represent the average for all items in the scale that the respondent answered.
Change in Beck Anxiety Inventory | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  The BAI is a 21-item self-report scale that assesses the severity of anxiety symptoms.
  Items are scored from 0 to 3 (0 = not at all, 3 = severe). Higher scores indicate greater levels of severity, and the ranges for anxiety levels are: 0-9 normal to minimal, 10-18 mild to moderate, 19-29 moderate to severe, and 30-63 severe. The BAI consists of two factors: somatic and cognitive.
Change in Respiratory Sinus Arrhythmia (RSA)- measured by PSG | Assessed at baseline (week 1), end of treatment (week 13), and 6-month follow-up (week 39)
  RSA is the phenomenon of an increased heart rate during inhalation and a decreased heart rate during exhalation. Since these fluctuations are controlled mainly by vagal influences on the heart, RSA serves as a reliable metric for measuring parasympathetic activity. RSA has been proven to be a reliable measure of emotion regulation and emotional responding in numerous studies.

CONTACTS AND LOCATIONS:
Locations (1):
- Stanford University, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No